CLINICAL TRIAL: NCT01063062
Title: A Single-arm, Open-label, Multicenter Study of Tocilizumab Monotherapy or in Combination With Methotrexate to Assess Safety and the Efficacy in Reducing Disease Activity in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Non-biologic DMARDs (PICTURE)
Brief Title: A Study With Tocilizumab [RoActemra/Actemra] Monotherapy or in Combination With Methotrexate in Patients With Rheumatoid Arthritis (PICTURE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22725
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

ARMS (1):
- tocilizumab (Experimental): Participants received an 8 mg/kg tocilizumab intravenous (IV) infusion once every 4 weeks for 24 weeks (6 infusions). Participants taking concomitant methotrexate (MTX) at Baseline remained on a stable dose as per standard of care at the Investigator's discretion.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Methotrexate

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenous infusion every 4 weeks.
Drug: Methotrexate — methotrexate as per standard of care in clinical practice.

SUMMARY:
This single-arm, open-label, multicenter study evaluated the safety and tolerability and the efficacy in reducing disease activity of tocilizumab [RoActemra/Actemra] as monotherapy or in combination with methotrexate in patients with active moderate to severe rheumatoid arthritis (RA). Patients were eligible to participate in this study if they are currently experiencing an inadequate response to a stable dose of a non-biologic disease-modifying antirheumatic drug (DMARD). Patients received 8 mg/kg tocilizumab [RoActemra/Actemra] as an intravenous infusion every 4 weeks for a total of 6 infusions. The anticipated time on study treatment was 24 weeks. The target sample size was 50-200 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age
* Moderate to severe rheumatoid arthritis (RA) for at least 6 months (defined as a Disease Activity Score (DAS28) > 3.2 at screening)
* Patients with active RA after more than 12 weeks of treatment with DMARDs
* Patients with inadequate response to a stable dose of non-biologic DMARD

Exclusion Criteria:

* Autoimmune disease other than RA. Patients with interstitial pulmonary fibrosis and able to tolerate methotrexate (MTX) and patients with Sjögren's Syndrome and RA are permitted
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following enrollment
* Prior history of or current inflammatory joint disease other than RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-02-28 (Actual); Primary Completion 2011-01-17 (Actual); Study Completion 2011-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Egypt (9):
  - Alexandria University Hospital; Rheumatology, Alexandria
  - Alexandria University, Alexandria
  - Banha Educational Hospital; Rheumatology, Banhā
  - Kasr El Ainy Hospital; Rheumatology, Cairo
  - Ain Shams University Hospital; Rheumatology, Cairo
  - Bab El Sheereya Hospital; Rheumatology, Cairo
  - El Hussein University Hospital; Rheumatology, Cairo
  - Kasr El Ainy Hospital, Cairo
  - Manial Specialized Hospital; Rheumatology, Cairo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 107 participants were enrolled from 11 centers in Egypt, 2 centers were prematurely terminated.
Pre-assignment Details: Patients in this 1 arm tocilizumab study were divided into 2 groups: tocilizumab monotherapy or tocilizumab plus methotrexate (patients taking disease-modifying antirheumatic drugs at Baseline who continued concomitant treatment with methotrexate as per standard of care at the investigator's discretion).
Groups:
- Tocilizumab: Participants received an 8 mg/kg tocilizumab intravenous (IV) infusion once every 4 weeks for 24 weeks (6 infusions).
- Tocilizumab + MTX: Participants received an 8 mg/kg tocilizumab intravenous (IV) infusion once every 4 weeks for 24 weeks (6 infusions). Participants taking concomitant methotrexate (MTX) at Baseline remained on a stable dose as per standard of care at the Investigator's discretion.
Period: Overall Study
Arm/Group | Tocilizumab | Tocilizumab + MTX
Started | 30 | 77
Received Study Drug | 29 | 76
Completed | 22 | 65
Not Completed | 8 | 12
Not completed — Patient withdrew consent | 0 | 1
Not completed — Adverse Event | 2 | 4
Not completed — Protocol Violation | 5 | 4
Not completed — Investigator's request | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Miscellaneous reason | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Tocilizumab Monotherapy: Participants received an 8 mg/kg tocilizumab intravenous (IV) infusion once every 4 weeks for 24 weeks (6 infusions).
- Total: Total of all reporting groups
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX | Total
Number analyzed (Participants) | 30 | 77 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.78 (12.47) | 41.76 (11.84) | 40.64 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 69 | 92
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Disease Activity Score 28 (DAS28) Low Disease Activity
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Low Disease Activity was defined as a DAS28 score of < 3.2.
Time Frame: Baseline to Week 24 (Weeks 4, 8, 12, 16, 20, 24)
Population: Intent-to-treat (ITT) population included all participants who received study drug and had at least 1 follow-up variable. Last observation carried forward was applied for missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
percentage of participants
  Week 4 | 27.59 | 18.42
  Week 8 | 34.48 | 40.79
  Week 12 | 34.48 | 38.16
  Week 16 | 44.83 | 47.37
  Week 20 | 62.07 | 57.89
  Week 24 | 58.62 | 59.21

2. Primary Outcome: Time to DAS28 Low Disease Activity
Description: Time to DAS28 Low Disease Activity was defined as the time in days from the first infusion of study drug to the achievement of a DAS28 Score <3.2 units. The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Low Disease Activity was defined as a DAS28 score of < 3.2.
Time Frame: 24 Weeks
Population: Intent-to-treat population included all participants who received at least one dose of study drug and had data for at least one follow-up variable available. Last observation carried forward.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Tocilizumab | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
days | 107.2 [84.57 to 129.78] | 100.2 [87.49 to 112.93]

3. Secondary Outcome: Percentage of Participants Achieving DAS28 Clinically Significant Improvement
Description: DAS28 Clinically Significant Improvement was defined as a DAS28 score reduction of at least 1.2 units from Baseline. The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24
Population: Intent-to-treat population included all participants who received study drug and had at least 1 follow-up variable. Last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
percentage of participants
  Week 4 | 62.07 | 73.68
  Week 8 | 75.86 | 86.84
  Week 12 | 75.86 | 90.79
  Week 16 | 79.31 | 92.11
  Week 20 | 82.76 | 90.79
  Week 24 | 86.20 | 96.10

4. Secondary Outcome: Time to DAS28 Clinically Significant Improvement
Description: Time to DAS28 Clinically Significant Improvement was the Time in days from the first infusion of study drug to the achievement of a DAS28 score reduction of at least 1.2 units. The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Low Disease Activity was defined as a DAS28 score of < 3.2.
Time Frame: 24 Weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
days | 59.9 [40.20 to 79.53] | 41.6 [34.51 to 48.76]

5. Secondary Outcome: Percentage of Participants Achieving DAS28 Remission
Description: DAS28 Remission was defined as a DAS28 score < 2.6 units. The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10.
Time Frame: Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
percentage of participants
  Week 4 | 17.24 | 9.21
  Week 8 | 31.03 | 23.68
  Week 12 | 31.03 | 27.63
  Week 16 | 34.48 | 34.21
  Week 20 | 41.38 | 40.79
  Week 24 | 48.28 | 40.79

6. Secondary Outcome: Time to DAS28 Remission
Description: Time to DAS28 Remission was the Time in days from the first infusion of study drug to the achievement of a DAS28 score < 2.6 units. The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10.
Time Frame: 24 Weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Tocilizumab | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
days | 115.9 [94.24 to 137.49] | 120.5 [108.38 to 132.57]

7. Secondary Outcome: Disease Activity Score 28 (DAS28)
Description: as for outcome 1
Time Frame: Weeks 4, 8, 12, 16, 20, 24
Population: Participants from the intent-to-treat population, all participants who received study drug and had at least 1 follow-up variable, with data available at the given time-point. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab | Tocilizumab + MTX
Number analyzed (Participants) | 25 | 75
score on a scale
  Week 4 (n=24,75) | 4.17 (1.45) | 4.48 (1.47)
  Week 8 | 3.72 (1.71) | 3.68 (1.60)
  Week 12 | 3.37 (1.62) | 3.54 (1.45)
  Week 16 | 3.25 (1.54) | 3.21 (1.43)
  Week 20 | 2.86 (1.50) | 3.11 (1.44)
  Week 24 | 2.51 (1.50) | 3.06 (1.51)

8. Secondary Outcome: C-Reactive Protein (CRP)
Description: Blood was collected for C-Reactive Protein (CRP), a test for inflammation, at Weeks 4, 8, 12, 16, 20 and 24 and was analyzed at a central laboratory. The serum concentration of CRP was measured in milligrams/deciliter (mg/dL).
Time Frame: Weeks 4, 8, 12, 16, 20, 24
Population: Participants from the intent-to-treat population, all participants who received study drug and had data for at least one follow-up variable, with data available for the given timepoint.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab | Tocilizumab + MTX
Number analyzed (Participants) | 25 | 75
mg/L
  Week 4 | 13.04 (24.90) | 12.28 (28.37)
  Week 8 (n=25,74) | 14.74 (35.74) | 6.24 (13.39)
  Week 12 | 9.35 (17.29) | 6.89 (15.84)
  Week 16 | 4.38 (9.98) | 3.87 (11.01)
  Week 20 | 7.92 (15.07) | 4.20 (12.11)
  Week 24 | 6.99 (13.64) | 3.82 (13.39)

9. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: Blood was collected for Erythrocyte Sedimentation Rate (ESR), a test to assess inflammation, at Weeks 4, 8, 12, 16, 20, 24 and was analyzed at a central laboratory. ESR was measured in millimeters/hour (mm/hr).
Time Frame: Weeks 4, 8, 12, 16, 20, 24
Population: Participants from the intent-to-treat population, all participants who received study drug and had at least 1 follow-up variable, with data available at the given time point. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 25 | 27
mm/hr
  Week 4 (n=24,27) | 21.08 (22.27) | 20.37 (25.66)
  Week 8 | 17.18 (21.54) | 13.79 (18.52)
  Week 12 | 14.12 (15.10) | 16.41 (22.25)
  Week 16 | 15.80 (23.65) | 13.88 (18.02)
  Week 20 | 16.32 (25.44) | 14.28 (20.42)
  Week 24 | 16.32 (22.43) | 16.40 (22.26)

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events. A SAE was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: 24 Weeks
Population: Safety population included all participants who received study drug and had post-dose safety data available.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
participants
  AEs | 29 | 76
  SAEs | 5 | 12

11. Secondary Outcome: Number of Participants With AE and SAE Related Discontinuation
Description: The number of participants who stopped using the study drug because of an AE or a SAE. An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events. A SAE was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: 24 Weeks
Population: Safety population included all participants who received study drug and had post-dose safety data available.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
participants
  Discontinuation due to AE | 8 | 7
  Discontinuation due to SAE | 5 | 6

12. Secondary Outcome: Number of Participants With Serious Infections
Description: A serious infection was an infection that qualified as a Serious Adverse Event (SAE). A SAE was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: 24 Weeks
Population: Safety population included all participants who received study drug and had post-dose safety data available.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
participants | 1 | 1

13. Secondary Outcome: Number of Participants With Elevated AST (SGOT) and ALT (SGPT)
Description: Blood was collected for aspartate aminotransferase (serum glutamic oxaloacetic transaminase) [AST/SGOT] and alanine aminotransferase (serum glutamic pyruvic transaminase) [ALT/SGPT], liver function tests, and were analyzed at a central laboratory. The number of participants with High AST (SGOT) or ALT (SGPT) levels at Week 24 is reported.
Time Frame: Week 24
Population: Participants from the safety population, all participants who received study drug and had at least 1 post-dose safety assessment, with data available for analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
participants
  ALT (SGPT) | 3 | 6
  AST (SGOT) | 3 | 8

14. Secondary Outcome: Number of Participants With Elevated Total Cholesterol According to ATPIII Guidelines
Description: Blood samples were collected for Total Cholesterol and were sent to a central laboratory for analysis. According to Adult Treatment Profile III (ATPIII) guidelines the Total Cholesterol level in milligram/deciliter (mg/dL) was categorized as: Desirable ( < 200), Borderline High (200- 239) or High (≥ 240). The number of participants categorized Borderline High or High at each time-point is reported.
Time Frame: Weeks 0 (Baseline), 4, 8, 12, 16, 20, 24
Population: Safety population included all participants who received study drug and had post-dose safety data available.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
participants
  Week 0 | 10 | 25
  Week 4 | 16 | 41
  Week 8 | 10 | 34
  Week 12 | 9 | 30
  Week 16 | 10 | 36
  Week 20 | 7 | 35
  Week 24 | 9 | 30

15. Secondary Outcome: Number of Participants With Elevated HDL Cholesterol According to ATPIII Guidelines
Description: Blood samples were collected for High Density Lipoprotein (HDL) Cholesterol and were sent to a central laboratory for analysis. According to Adult Treatment Profile III (ATPIII) guidelines the HDL Total Cholesterol level in milligram/deciliter (mg/dL) was categorized as: Low (< 40) or High (≥ 60). The number of participants with category High at each time-point is reported.
Time Frame: Weeks 0 (Baseline), 4, 8, 12, 16, 20, 24
Population: Safety population included all participants who received study drug and had post-dose safety data available.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 75
participants
  Week 0 | 4 | 20
  Week 4 | 10 | 34
  Week 8 | 2 | 26
  Week 12 | 6 | 22
  Week 16 | 5 | 19
  Week 20 | 2 | 20
  Week 24 | 5 | 20

16. Secondary Outcome: Number of Participants With Elevated LDL Cholesterol According to ATPIII Guidelines
Description: Blood samples were collected for Low Density Lipoprotein (LDL) Cholesterol and were sent to a central laboratory for analysis. According to Adult Treatment Profile III (ATPIII) guidelines the LDL Cholesterol level in milligram/deciliter (mg/dL) was categorized as: Optimal (< 100), Near Optimal/Above Optimal (100- 129), Borderline High (130- 159), High (160-189) or Very High (≥ 190). The number of participants categorized Borderline High, High or Very High at each time-point is reported.
Time Frame: Weeks 0 (Baseline), 4, 8, 12, 16, 20, 24
Population: Safety population included all participants who received study drug and had post-dose safety data available.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
participants
  Week 0 | 9 | 24
  Week 4 | 11 | 35
  Week 8 | 7 | 21
  Week 12 | 8 | 27
  Week 16 | 9 | 31
  Week 20 | 7 | 33
  Week 24 | 8 | 29

17. Secondary Outcome: Number of Participants With Elevated Triglyceride According to ATPIII Guidelines
Description: Blood samples were collected for Triglyceride and were sent to a central laboratory for analysis. According to Adult Treatment Profile III (ATPIII) guidelines the Triglyceride level in milligram/deciliter (mg/dL) was categorized as: Normal (< 150), Borderline High (150- 199), High (200- 499) or Very High (≥ 500). The number of participants categorized Borderline High, High or Very High at each time-point is reported.
Time Frame: Weeks 0 (Baseline), 4, 8, 12, 16, 20, 24
Population: Safety population included all participants who received study drug and had post-dose safety data available.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Number analyzed (Participants) | 29 | 76
participants
  Week 0 | 4 | 7
  Week 4 | 6 | 15
  Week 8 | 4 | 12
  Week 12 | 5 | 15
  Week 16 | 6 | 15
  Week 20 | 8 | 16
  Week 24 | 6 | 16

ADVERSE EVENTS:
Description: Safety population included all participants who received study drug and had post-dose safety data available.
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + MTX
Serious Adverse Events (participants affected / at risk) | 5/29 | 12/76
Other Adverse Events (participants affected / at risk) | 29/29 | 76/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Monotherapy (N=29) | Tocilizumab + MTX (N=76)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Viremia (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Gangrene (Infections and infestations) | 1 | 0
Hepatitis fulminant (Hepatobiliary disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Chest pain (General disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Monotherapy (N=29) | Tocilizumab + MTX (N=76)
Anaemia (Blood and lymphatic system disorders) | 10 | 24
Anisocytosis (Blood and lymphatic system disorders) | 1 | 5
Hypochromic anaemia (Blood and lymphatic system disorders) | 4 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 9
Leukopenia (Blood and lymphatic system disorders) | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 5 | 17
Vertigo (Ear and labyrinth disorders) | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Gastritis (Gastrointestinal disorders) | 3 | 2
Gingivitis (Gastrointestinal disorders) | 2 | 3
Fatigue (General disorders) | 2 | 1
Generalised oedema (General disorders) | 0 | 5
Oedema (General disorders) | 2 | 5
Oedema peripheral (General disorders) | 0 | 5
Pain (General disorders) | 4 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 4
Nasopharyngitis (Infections and infestations) | 3 | 5
Alanine aminotransferase increased (Investigations) | 5 | 17
Aspartate aminotransferase increased (Investigations) | 5 | 19
Bilirubin conjugated increased (Investigations) | 5 | 10
Blood albumin increased (Investigations) | 2 | 5
Blood alkaline phosphatase decreased (Investigations) | 2 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Blood bilirubin increased (Investigations) | 2 | 7
Blood bilirubin unconjugated increased (Investigations) | 2 | 3
Blood calcium decreased (Investigations) | 12 | 29
Blood chloride decreased (Investigations) | 6 | 13
Blood chloride increased (Investigations) | 16 | 55
Blood cholesterol (Investigations) | 2 | 3
Blood cholesterol increased (Investigations) | 12 | 42
Blood creatinine decreased (Investigations) | 4 | 5
Blood creatinine increased (Investigations) | 2 | 3
Blood phosphorus increased (Investigations) | 4 | 9
Blood potassium decreased (Investigations) | 3 | 2
Blood potassium increased (Investigations) | 2 | 5
Blood pressure decreased (Investigations) | 0 | 4
Blood pressure diastolic increased (Investigations) | 3 | 9
Blood pressure increased (Investigations) | 1 | 10
Blood sodium increased (Investigations) | 11 | 28
Blood triglycerides increased (Investigations) | 9 | 28
Blood urea increased (Investigations) | 3 | 9
Blood uric acid increased (Investigations) | 4 | 15
Haematocrit decreased (Investigations) | 7 | 23
Haemoglobin decreased (Investigations) | 8 | 15
Hepatic enzyme increased (Investigations) | 7 | 14
Low density lipoprotein (Investigations) | 1 | 4
Low density lipoprotein increased (Investigations) | 18 | 59
Mean cell haemoglobin concentration decreased (Investigations) | 4 | 2
Mean cell haemoglobin decreased (Investigations) | 7 | 7
Mean cell volume decreased (Investigations) | 4 | 5
Neutrophil count decreased (Investigations) | 4 | 7
Platelet count decreased (Investigations) | 0 | 6
Red blood cell count decreased (Investigations) | 5 | 18
Red blood cell count increased (Investigations) | 5 | 9
Red cell distribution width increased (Investigations) | 6 | 16
Very low density lipoprotein increased (Investigations) | 3 | 15
White blood cell count decreased (Investigations) | 3 | 10
White blood cell count increased (Investigations) | 4 | 9
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 9
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 | 15
Hypernatraemia (Metabolism and nutrition disorders) | 6 | 14
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 21
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 3
Headache (Nervous system disorders) | 3 | 10
Somnolence (Nervous system disorders) | 0 | 4
Renal colic (Renal and urinary disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 4 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 4
Hypertension (Vascular disorders) | 2 | 13
Hypotension (Vascular disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.